CLINICAL TRIAL: NCT05057819
Title: Randomized, Double-blind, Placebo-controlled Crossover Trial Assessing the Impact of the SGLT2 Inhibitor Empagliflozin on Postprandial Hypoglycaemia After Gastric Bypass
Brief Title: Investigating the Impact of the SGLT2 Inhibitor Empagliflozin on Postprandial Hypoglycaemia After Gastric Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DEEP-Empa
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Dumping Syndrome; Hypoglycemia, Reactive
MeSH Terms: conditions — Dumping Syndrome; Hypoglycemia | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, crossover trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin first, Placebo second (Experimental): Oral empagliflozin 25 mg daily in the morning for 20 days, followed by oral placebo (daily in the morning) for 20 days after a wash-out period of 2-6 weeks
  Interventions: Drug: Empagliflozin 25 MG; Drug: Placebo
- Placebo first, Empagliflozin second (Placebo Comparator): Oral placebo (daily in the morning) for 20 days, followed by oral empagliflozin 25 mg daily in the morning for 20 days after a wash-out period of 2-6 weeks
  Interventions: Drug: Empagliflozin 25 MG; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Treatment naive patients with bariatric bypass surgery will be given oral empagliflozin 25mg once daily for 20 days
Drug: Placebo — Treatment naive patients with bariatric bypass surgery will be given oral placebo once daily for 20 days

SUMMARY:
Bariatric surgery is an effective anti-obesity treatment providing durable weight loss and profound beneficial effects on glucose metabolism. However, bariatric surgery also comes with an increased risk for a late metabolic complication known as postbariatric hypoglycaemia (PBH). The condition presents with hypoglycaemic episodes 1-3 hours after meals and develops one to several years after bariatric surgery, mainly gastric bypass. PBH affects approximately 30% of patients without preexisting diabetes. For a subset of patients, hypoglycaemia-associated impairment of daily living and social functioning are commonly observed. The underlying mechanisms of PBH are multifactorial. It is considered that inadequately high insulin secretion caused by both accelerated glucose absorption from the gut and increased insulinotropic hormones such as GLP-1 are important pathophysiologic mechanisms. Empagliflozin, a sodium-glucose cotransporter 2 (SGLT2) inhibitor reduces glucose exposure by increasing urinary glucose excretion. In a pilot study, a single dose of 10mg of empagliflozin taken before a mixed meal reduced the risk of PBH by 74%. Both, postprandial glucose and insulin exposure were significantly lower with empagliflozin vs. placebo, which makes Empagliflozin a potential treatment for PBH. In this study, treatment naïve patients will be randomized to receive either oral empagliflozin 25 mg daily in the morning for 20 days, followed by 2-6 weeks wash out and 20 days placebo once daily in the morning, or the reverse sequence. Urine and blood analysis will be performed as detailed in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age 18 years or older
* Gastric bypass surgery ≥1 year ago
* Biochemically confirmed postprandial hypoglycaemia (plasma or sensor glucose <3.0mmol/l) within the past three months

Exclusion Criteria:

* Diabetes on anti-diabetic treatment (insulin and/or non-insulin agents)
* Genito-urinary infection, if not treated successfully
* Chronic kidney disease (defined as CKD-EPI eGFR < 60 mL/min per 1.73 m2 body surface area)
* Pregnant and lactating women (urine pregnancy test to be performed for women of childbearing potential [defined as women who are not surgically sterilized/ hysterectomized, and/ or who are postmenopausal for less than 12 months]) or women of childbearing potential that refuse to use an effective contraceptive method [birth control pill or intrauterine device (IUD)]).
* Inability to understand and follow the protocol
* Known allergy to the study drug
* Participation in another interventional clinical trial overlapping with the current trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Amplitude of change in plasma glucose (difference between peak and nadir plasma glucose concentration in mmol/L) during the mixed meal test. | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, the amplitude of plasma glucose (difference between peak and nadir plasma glucose concentration in mmol/L) will be measured.

SECONDARY OUTCOMES:
Mean amplitude of glucose excursion (MAGE) based on CGM glucose | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo (i.e. aggregated measures of the outcome will be calculated for each period). The first 3 days of data of each period will be discarded.
  During the intake of empagliflozin and placebo, participants will wear a continuous glucose monitoring device. After V1 and V2, CGM data will be extracted and analysed. MAGE will be calculated based on CGM data obtained during each observation period.
Mean coefficient of variability based on CGM glucose | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo (i.e. aggregated measures of the outcome will be calculated for each period). The first 3 days of data of each period will be discarded.
  During the intake of empagliflozin and placebo, participants will wear a continuous glucose monitoring device. After V1 and V2, CGM data will be extracted and analysed. The mean coefficient of variability will be calculated based on CGM data obtained during each observation period.
Peak plasma glucose during mixed meal test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, the peak of plasma glucose (in mmol/L) will be documented.
Percent time spent with CGM glucose >10.0mmol/L | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo (i.e. aggregated measures of the outcome will be calculated for each period). The first 3 days of data of each period will be discarded.
  During the intake of empagliflozin and placebo, participants will wear a continuous glucose monitoring device. After V1 and V2, CGM data will be extracted and analysed. Percent time spent with CGM glucose >10.0mmol/L will be calculated based on CGM data obtained during each observation period.
Proportion of participants experiencing hypoglycaemia (defined as plasma glucose<3.0mmol/L) during the mixed meal tolerance test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, the proportion of participants experiencing hypoglycaemia (defined as plasma glucose<3.0mmol/L) will be documented.
Nadir plasma glucose during mixed meal test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, the nadir of plasma glucose (in mmol/L) will be documented.
Percent time spent with CGM glucose <3.0mmol/L | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo (i.e. aggregated measures of the outcome will be calculated for each period). The first 3 days of data of each period will be discarded.
  During the intake of empagliflozin and placebo, participants will wear a continuous glucose monitoring device. After V1 and V2, CGM data will be extracted and analysed. Percent time spent with CGM glucose <3.0mmol/L will be calculated based on CGM data obtained during each observation period.
Percent time spent with CGM glucose <2.8mmol/L | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo (i.e. aggregated measures of the outcome will be calculated for each period). The first 3 days of data of each period will be discarded.
  During the intake of empagliflozin and placebo, participants will wear a continuous glucose monitoring device. After V1 and V2, CGM data will be extracted and analysed. Percent time spent with CGM glucose <2.8mmol/L will be calculated based on CGM data obtained during each observation period.
Frequency of postprandial symptoms based on a modified Edinburgh Hypoglycaemia | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo.
  During the intake of empagliflozin and placebo, participants will report postprandial symptoms in an electronic event diary. The frequency of postprandial symptoms, based on a modified Edinburgh Hypoglycaemia Symptom Scale, will be documented.

OTHER OUTCOMES:
Measures of beta-cell function using the oral minimal model method calculated using data from the mixed-meal test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. Measures of beta-cell function will be calculated using the oral minimal model method with data from the mixed-meal test.
Measures of insulin sensitivity using the oral minimal model method calculated using data from the mixed-meal test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. Measures of insulin sensitivity will be calculated using the oral minimal model method with data from the mixed-meal test.
Measures of first-pass hepatic insulin extraction using the oral minimal model method calculated using data from the mixed-meal test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. Measures of first-pass hepatic insulin extraction will be calculated using the oral minimal model method with data from the mixed-meal test.
Average daily meal frequency (meals>30g/24h and meals <30g/24h) assessed during the treatment periods | The outcome will be calculated from day 1 to day 20 of intake of IMP/Placebo.
  During the intake of empagliflozin and placebo, participants will report meals in an electronic event diary. Average daily meal frequency per 24 hours will be calculated.
Total amount of daily excreted glucose (g/24h) measured in the 24h urine collection | The outcome will be assessed during the day before the experimental visit.
  The participants will collect a 24-hours urine sample on the day before the mixed meal test. Total amount of daily excreted glucose (in grams per 24 hours) will be calculated.
Glucagon response during the mixed-meal test (incremental AUC from 0 to 120min following meal ingestion) | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, the plasma glucagon concentrations will be measured.
Insulin response during the mixed-meal test (incremental AUC from 0 to 120min following meal ingestion) | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, the plasma insulin concentrations will be measured.
Ketone levels (3-beta-hydroxybutyrate) during the mixed-meal test | The outcome will be assessed during the mixed-meal test on the day of the experimental visit at the end of each study period (day 20-24 of the respective study period).
  On day 20 of the intake of either empagliflozin or placebo, participants undergo a mixed meal test. During the test, ketone levels (3-beta-hydroxybutyrate) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD/PhD, Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital and University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After study completion, 10 years
Access Criteria: After written inquiry and approval by the principal investigator

REFERENCES:
- [Derived] Ferreira A, Schonenberger KA, Potoczna N, Vogt A, Gerber PA, Zehetner J, Giachino D, Nett P, Gawinecka J, Cossu L, Fuster DG, Dalla Man C, Facchinetti A, Melmer A, Nakas CT, Hepprich M, Donath MY, Herzig D, Bally L. Randomized, Double-Blind, Placebo-Controlled Crossover Trial of Once Daily Empagliflozin 25 mg for the Treatment of Postprandial Hypoglycemia After Roux-en-Y Gastric Bypass. Diabetes Technol Ther. 2023 Jul;25(7):467-475. doi: 10.1089/dia.2023.0036. Epub 2023 Jun 5. PMID 37093196
- [Derived] Ferreira A, Emara AFA, Herzig D, Melmer A, Vogt AP, Nakas CT, Facchinetti A, Dalla Man C, Bally L. Study protocol for a randomised, double-blind, placebo-controlled crossover trial assessing the impact of the SGLT2 inhibitor empagliflozin on postprandial hypoglycaemia after gastric bypass. BMJ Open. 2022 Sep 19;12(9):e060668. doi: 10.1136/bmjopen-2021-060668. PMID 36123073